CLINICAL TRIAL: NCT02809794
Title: CPAP In-home Assessment Australia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA175
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational CPAP device (Experimental): Fisher & Paykel Healthcare CPAP Device
  Interventions: Device: Fisher & Paykel Healthcare CPAP Device

INTERVENTIONS:
Device: Fisher & Paykel Healthcare CPAP Device — Fisher & Paykel Healthcare CPAP Device

SUMMARY:
The study is to evaluate the product reliability, therapy effectiveness and user feedback of a Continuous Positive Airway Pressure (CPAP) device in-home for up to 6 months.

DETAILED DESCRIPTION:
Existing and Naïve CPAP users will be recruited into a 6 month in-home study Participants will attend 5 study visits at day 0, 7, 30, 60 and 180. Outcome of the clinical investigation include downloadable device data reports, device error reports and participants perception questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over.
* Diagnosed with OSA by a practicing physician and prescribed Positive Airway Pressure (PAP) therapy.

Exclusion Criteria:

* Persons contraindicated for Continuous Positive Airway Pressure (CPAP) therapy.
* Persons with other significant sleep disorder(s) (e.g. periodic leg movements, insomnia, central sleep apnea).
* Persons with obesity hypoventilation syndrome or congestive heart failure.
* Persons that require supplemental oxygen with their CPAP device.
* Persons with implanted electronic medical devices (e.g. cardiac pacemakers).
* Persons who are pregnant or think they might be pregnant.
* Persons whose primary language is other than English.
* Persons in existing dependent or unequal relationships with any member of the research team, the researcher(s) and/or the person undertaking the recruitment/consent process.
* Persons highly dependent on medical care.
* People with cognitive impairment, an intellectual disability or a mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI), measured as number of events/hour | 6 months
  Obtained from the device
Log of safety-related events, measured as number of safety-related faults | 6 months
  Obtained from the device
Machine reported faults, measured as number of machine faults | 6 months
  Obtained from the device
Participant reported faults, measured as number of participant complaints | 6 months
  Obtained from the follow up visits

SECONDARY OUTCOMES:
Perception of the device, measured through questionnaire | 6 months
  Impression of the device during the follow up visits

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Sleep Matters, Bulleen, Victoria
  - Sleep & Snore Solutions, Bunbury, Western Australia
  - St John of God Midland Public Hospital, Midland, Western Australia